CLINICAL TRIAL: NCT07115225
Title: Predictive Validity of an Upper Extremity Physical Performance Test Battery in Patients After Shoulder Dislocation: a Prospective Study
Brief Title: Validation of an Upper Extremity Physical Performance Test Battery in Patients After Shoulder Dislocation
Acronym: VAL_PPT_P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: AZ Monica Campus Antwerpen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2024-0629
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Return to Sport; Shoulder Dislocation or Subluxation
MeSH Terms: conditions — Shoulder Dislocation; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients after shoulder stabilization procedure (Latarjet or Bankart procedure) (Experimental): Patients who underwent shoulder stabilization surgery (Latarjet or Bankart procedure) between the ages of 16 and 55 years old
  Interventions: Other: Analytical test - Shoulder Range of Motion (ROM); Other: Analytical test - Shoulder Strength; Other: Modified-Athletic Shoulder Test (M-AST); Other: Physical performance test - Unilateral Seated Shot-Put Test (USSPT); Other: Physical performance test - modified-Closed Kinetic Chain Upper Extremity Stability Test (m-CKCUEST); Other: Supine moving apprehension test (SMAT); Other: Physical performance test - Posterior shoulder endurance test (PSET); Other: Patient-reported outcome measure - The Shoulder Instability-Return to Sport after Injury (SIRSI); Other: Patient-reported outcome measure - Numeric Pain Rating Scale (NPRS); Other: Modified Tampa-Scale of Kinesiophobia for Anterior Shoulder Instability (TSK-SI)

INTERVENTIONS:
Other: Analytical test - Shoulder Range of Motion (ROM) — Passive external rotation in supine position with arm in 90° abduction - passive internal rotation in supine position with arm in 90° abduction.
Other: Analytical test - Shoulder Strength — Shoulder external rotation and internal rotation measured with a hand held dynanometer in supine lying
Other: Modified-Athletic Shoulder Test (M-AST) — Shoulder strength in the antero-posterior plane measured with a hand held dynanometer in prone lying
Other: Physical performance test - Unilateral Seated Shot-Put Test (USSPT) — Set up requires that the subject is placed in a seated position (knees bent at 90° degrees) with their back against the wall, and a 3 kg medicine ball held at height of the shoulder. When ready, the subject will perform a shot put motion to push the medicine ball as far as possible in a horizontal direction. The average of three trials is recorded for each arm.
Other: Physical performance test - modified-Closed Kinetic Chain Upper Extremity Stability Test (m-CKCUEST) — The test is performed in a push-up position with the hands one half-arm span apart on strips of athletic tape. The person reaches with alternating hands across the body to touch the piece of tape under the opposing hand. The number of cross-body touches performed in 15 seconds is recorded. In total, three 15-s test trials were performed, with 45 s rest between each trial.
Other: Supine moving apprehension test (SMAT) — The beginning position of the participant is lying in a supine position while holding the weight just over their chest. Participants move their shoulder to 135° of abduction with the elbow extended, then returning to the starting position, and immediately move their shoulder to 180° of abduction with the elbow fully extended and finally return to the starting position. This cycle is repeated as much as possible for 1 minute.
Other: Physical performance test - Posterior shoulder endurance test (PSET) — The participant is positioned prone, with the test shoulder off the table and the arm in 90° of horizontal abduction, the point at which the participant is to hold the arm as long as possible until fatigue. The participant holds a weight equal to 2% of his body weight (rounded to the nearest 0.5 kg).
Other: Patient-reported outcome measure - The Shoulder Instability-Return to Sport after Injury (SIRSI) — Psycho-social questionnaire assessing the psychological readiness of athletes to return to sport following traumatic shoulder instability and conservative or surgical management. The SIRSI includes 12 questions with an 11-point Likert scale in the form of blocks to be ticked from 0 to 10. The total score is equal to the sum of the values of the 12 responses then determined in relation to 100 to obtain a percentage. High scores correspond to a positive psychological response.
Other: Patient-reported outcome measure - Numeric Pain Rating Scale (NPRS) — Patient's shoulder pain will be measured using an 11-point NRS, with a minimum value of zero ("no pain") and a maximum score of 10 ("the worst pain possible")
Other: Modified Tampa-Scale of Kinesiophobia for Anterior Shoulder Instability (TSK-SI) — modified Tampa Scale of Kinesiophobia (TSK) to make it suitable for application in patients with anterior shoulder instability. The TSK-SI contains 18 items and the total score can range from 18 to 72, with 18 being the "best" score (no fear of movement/kinesiophobia) and 72 being the "worst" score (severe fear of movement/kinesiophobia)

SUMMARY:
The goal of this exploratory prospective study is to determine if an upper extremity test battery, comprised of physical performance tests, analytical tests and patient-reported outcome measures, can predict successful return to sports and quality of life in athletes (age 16-55) after shoulder dislocation.

The main research questions are:

* Can an Upper Extremity Physical Performance Test Battery predict successful return to sports (= return to pre-injury sports level) in athletes after shoulder stabilization procedure
* Can an Upper Extremity Physical Performance Test Battery predict the quality of life in athletes after shoulder stabilization procedure

Participants will:

* Fill out questionnaires pre-operatively
* Fill out the SIRSI questionnaire throughout the rehabilitation
* Undergo a testing battery in the return to sport phase, including physical performance tests, analytical tests and patient-reported outcome measures
* Fill out questionnaires every 3 months after return to sports, up to 1 year.

DETAILED DESCRIPTION:
After enrollment, athletes will be asked about their injury history, and demographic information will also be collected, including gender, age, athlete experience, and sports level. During rehabilitation (duration: typically between 3 and 6 months), the participant will be given a monthly questionnaire that surveys their rehabilitation progress. At the time they return to sport (after green light by orthopaedic surgeon and physiotherapist), they are tested once with the test battery (physical performance tests, analytical tests and patient-reported outcome measures). Patients will be tested as close as possible to the actual return to sport timing. Following, they are monitored for another year with questionnaires, every 3 months, that survey their pain, current level of competition, quality of life, confidence in the shoulder and possible re-injuries. This way, the included participants will be monitored for +- 18 months (duration of rehabilitation + 1 year follow-up after return to sport).

ELIGIBILITY:
Inclusion Criteria:

* Practising sports with moderate to high demand on the shoulder (based on Degree of Shoulder Involvement in Sport (DOSIS) scale), minimal weekly 3 hours
* Shoulder instability event (anterior direction)
* Healthy contralateral shoulder
* Completion of the postoperative rehabilitation protocol

Exclusion Criteria:

* Other upper limb pathologies/ associated injuries: e.g. posterior instability, or rotator cuff tear,...
* Being pregnant
* No intention to return to pre-injury sport

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Patient Outcome for Return to Sports (SPORTS) score | 3 months, 6 months, 9 months, 12 months post-return to sport
  Subjective Patient Outcome for Return to Sports (SPORTS) score is a single-item scale that measures athletes' ability to return to their preinjury sport based on effort and performance. It is scored on a 10-point scale with 0 points allocated to the patient who does not resume the same sport and 10 points to the patient who is able to perform, without pain, the same sport, at same level of effort and performance as before the onset of his/her impairment.
Western Ontario Shoulder Instability Index (WOSI) | pre-operatively; in return to sport phase; 3 months, 6 months, 9 months, 12 months post-return to sport
  The WOSI score questionnaire is a tool designed for self-assessment of shoulder function for patients with shoulder instability. It consists of four subscales with a total of 21 items. Each question in this version is scaled on a Numerical Rating Scale from 0 (best) to 10 (worst), with the WOSI score ranging from 0 (highest shoulder-related quality of life) to 210 (worst shoulder-related quality of life).

SECONDARY OUTCOMES:
Re-injury | 3 months, 6 months, 9 months, 12 months post-return to sport
  The questionnaire will capture re-injuries and subsequent injuries within 12 months after return to sport

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - AZ Monica, Deurne - Orthopedie, Antwerp
  - Department of rehabilitation sciences, Ghent university, Ghent

IPD SHARING:
Plan to Share IPD: Undecided